CLINICAL TRIAL: NCT04419428
Title: A40 EFL Registry: A Multicenter Prospective Study to Determine the Role of Expiratory Flow Limitation (EFL) in Patients With Chronic Obstructive Pulmonary Disease (COPD) Receiving Home Mechanical Ventilation
Brief Title: A40 Expiratory Flow Limitation Registry
Status: Withdrawn | Type: Observational
Why Stopped: Philips placed the study on hold in August 2022 due to the awareness of a potential device functionality issue. Philips has shifted business priorities and has decided to cancel the trial.
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: SRC_HRC_VectorEUReg_2019_10820
Record Dates: First submitted 2020-05-14; First posted 2020-06-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Noninvasive ventilation; Daytime Hypercapnia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: BiPAP A40 Expiratory Flow Limitation (EFL) — All participants in the observational registry will be using the BiPAP A40 EFL noninvasive ventilator as part of standard of care and will be participating in the same follows up and data collection. The BiPAP A-40 EFL ventilator is intended to provide non-invasive ventilatory support to treat adult patients with Respiratory Insufficiency with the primary cause being COPD. It is intended to be used within the home, institution/hospital, and diagnostic laboratory environments.

SUMMARY:
This prospective observational multicenter registry study will include adults greater than 40 years old, diagnosed with chronic obstructive pulmonary disease, requiring home noninvasive ventilation as part of standard medical care. For the purposes of this study, chronic obstructive pulmonary disease is defined as chronic respiratory failure consisting of historical spirometry vales (FEV1 <60% predicted and FEV1/VC < 0.7) and chronic increased daytime carbon dioxide levels greater than 6.0 kPa or 45 mmHg. In addition, participants diagnosed with major organ system diseases or obstructive sleep apnea will be excluded. At least 100 men and women who consent and meet the inclusion/exclusion criteria will be asked to participate. The anticipated study duration will be 6 months. The study will involve an initial visit for the standard of care initiation of home noninvasive ventilation. At this time, potential participants will be screened for participation. If eligible once consented, medical history will be collected and baseline questionnaires related to their respiratory disease will be completed. The registry study will include 6 month of home use of the noninvasive ventilator using the BiPAP A40 EFL device. Study staff will reach out to participants on a monthly basis to review any issues, medication changes, unscheduled visits, and device data download. Additional phone calls and or visits may occur on an as needed basis if issues arise. The final visit will be an in facility visit. The primary endpoint will be the overall prevalence of Expiratory Flow Limitation (EFL) in ventilated hypercapnic COPD patients, as defined as the percentage participants exhibiting a DeltaXrs value greater than or equal to 2.8 during one or more nights of therapy.

DETAILED DESCRIPTION:
Prospective observational multicenter registry study for chronic obstructive pulmonary disease patients who require noninvasive ventilation in the home setting as part of standard medical care. The registry includes one in person screening or baseline visit, monthly follow-up phone calls (monitoring for medication changes, unscheduled visits and adverse events) and device data downloads, and a final in person study visit.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Forced Expiratory Volume (FEV1) < 60% predicted
* Forced Expiratory Volume (FEV1) / Vital Capacity (VC) ratio < 0.7
* Greater than 40 years old
* Chronic hypercapnia (daytime carbon dioxide level PaCO2 > 6.0 kPa)
* No clinical diagnosis of Obstructive Sleep Apnea
* Smoking history > 10 pack year
* Body mass index (BMI) ≤ 35kg/m2

Exclusion Criteria:

* Hypercapnic respiratory acidosis defined as pH (measure of hydrogen ion, measure of the acidity or alkalinity of a fluid) <7.35
* Acute coronary syndrome and unstable angina
* Cognitive impairment that would prevent informed consent into the trial and/or inability to comply with the protocol
* Patients undergoing renal replacement therapy
* Patients with serious comorbidities confirming prognosis likely to be less than 12-months
* Pregnancy
* Congestive Heart Failure (CHF) with ejection fraction (EF) less than 45% determined by Echo if available

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female adults greater than 40 years old, diagnosed with chronic obstructive pulmonary disease, requiring home noninvasive ventilation as part of standard medical care. For the purposes of this study, chronic obstructive pulmonary disease is defined as chronic respiratory failure consisting of historical spirometry vales (FEV1 <60% predicted and FEV1/VC < 0.7) and chronic increased daytime carbon dioxide levels greater than 6.0 kPa or 45 mmHg. In addition, participants diagnosed with major organ system diseases or obstructive sleep apnea will be excluded. At least 100 men and women who consent and meet the inclusion/exclusion criteria will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Screening Expiratory flow limitation | Screening
  Percentage of participants exhibiting an expiratory flow limitation (Delta Xrs value) greater than or equal to 2.8 at the time of screening.
Expiratory flow limitation post therapy | 6 months
  Percentage of participants exhibiting an expiratory flow limitation (Delta Xrs value) greater than or equal to 2.8 during one of more nights of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Polkey, MD, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No